CLINICAL TRIAL: NCT01312545
Title: Comparison of Exposure Rate Between Local Made and Imported Porous Polyethylene Orbital Implant for Enucleation in Thailand: A Randomized, Equivalence Controlled Trial and Multicenter Study
Brief Title: Comparison of Local Made and Imported Porous Polyethylene Orbital Implant for Enucleation in Thailand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mettapracharak Hospital (Other Government)
Collaborators: Thailand Research Fund (Other); Prince of Songkla University (Other); National Research Council of Thailand (Other Government); National Science and Technology Development Agency, Thailand (Other Government)
Responsible Party: Principal Investigator, Dr. Sunisa Sintuwong, Dr., Mettapracharak Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MEC1/2011
Record Dates: First submitted 2011-03-07; First posted 2011-03-10 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Phthisis Bulbi
Keywords: orbital implant; evisceration; economic; polyethylene; porous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- local made implant (3DP) (Experimental): Enucleation and local made implant (3DP) insertion
  Interventions: Device: 3DP
- imported implant (Medpor) (Experimental): Enucleation and imported implant (Medpor) insertion
  Interventions: Device: Medpor

INTERVENTIONS:
Device: 3DP — intervention involving local made implant with different fabricating technique-3-dimensional printing (3DP) technique.
  Arms: local made implant (3DP)
Device: Medpor — commercial porous polyethylene
  Arms: imported implant (Medpor)

SUMMARY:
This study wants to compare between two types of implants in enucleation. Both of them are made from porous polyethylene but have different fabricating techniques. The investigators chose an exposure rate as a main outcome because the investigators think it is the most important outcome for the surgeons. The study hypothesis is: Is the exposure rate of a local-made polyethylene orbital implant the same as an imported one?

DETAILED DESCRIPTION:
Sample size assessment

* The sample size was calculated by using an equivalence formula. From a literature and our own experiences, the success rate for Medpor and 3DP were 92% and 94% respectively, the difference (D) of the success rate between two groups was 10% and assuming a 15% of drop out rate.
* Then allocation sequence was generated by a computerized program, using block of six with varying block size.

Data management

* All definition of data, recruiting techniques, data collection techniques and data management flow were mentioned in the SOP.
* After double entry technique, each case record form from each site will be sent via DataFax system to the data center at Center of Excellence for Biomedical and Public Health Informatics (BIOPHICS), Thailand.
* Then data will be validated, analyzed and reported by staff at BIOPHICS.

Plan for missing data

* by adding a drop out rate to the sample size calculation.
* by choosing the right patients. Actually, Thai patients have good co-operation especially in surgical research.

Statistical analysis

- Intention to treat and per protocol model would be used to see the difference between two types of implants in this project.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of phthisis bulbi, painful blindness, intraocular tumor without metastasis and severe ruptured eyeball
* Must speak and understand Thai language well
* Must have good consciousness

Exclusion Criteria:

* Has a history of prior enucleation or evisceration
* Cannot follow up for at least one year
* Has recent eye infection within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2011-03; Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Exposure rate | From date of surgery until the date of first exposure, assessed up to 12 months
  Exposure was defined as the separation of tissue over the anterior surface of an implant.

SECONDARY OUTCOMES:
Infection rate | From date of surgery until the date of first infection, assessed up to 12 months
  Infection was defined as the presence of pus or abscess at or around an implant. It can be diagnosed clinically or confirmed by the histopathology report after explantation.

CONTACTS AND LOCATIONS:
Overall Officials: Sunisa Sintuwong, MD,MPPM,MSc, Principal Investigator — Mettapracharak (Wat Rai Khing) Hospital
Locations (1):
- Mettapracharak Eye Center, Mettapracharak (Wat Rai Khing) Hospital, Sam Phran, Changwat Nakhon Pathom, Thailand

IPD SHARING:
Plan to Share IPD: No